CLINICAL TRIAL: NCT04198363
Title: A Randomized Double-Blind, Phase 3 Study to Evaluate the Efficacy and Safety of Bismuth-Containing Quadruple Therapy With Oral TAK-438 20 mg Compared to Esomeprazole 20 mg Twice Daily in Subjects With Helicobacter Pylori Infection
Brief Title: A Study to Evaluate the Efficacy and Safety of Bismuth-Containing Quadruple Therapy With Oral Vonoprazan (TAK-438) 20 mg Compared to Esomeprazole 20 mg Twice Daily in Paticipants With Helicobacter Pylori Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vonoprazan-3002
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2022-10

CONDITIONS: Helicobacter Pylori
Keywords: Drug Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Clarithromycin; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan 20 mg (Experimental): Vonoprazan 20 mg, tablets, orally, twice daily given in combination with bismuth containing quadruple therapy (amoxicillin 1 gm, capsules, clarithromycin 500 mg, tablets, and bismuth potassium citrate 600 mg) orally, twice daily for up to 2 weeks.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Bismuth Potassium citrate
- Esomeprazole 20 mg (Active Comparator): Esomeprazole 20 mg, tablets, orally, twice daily given in combination with bismuth containing quadruple therapy (amoxicillin 1 gm, capsules, clarithromycin 500 mg, tablets, and bismuth potassium citrate 600 mg) orally, twice daily for up to 2 weeks.
  Interventions: Drug: Amoxicillin; Drug: Clarithromycin; Drug: Bismuth Potassium citrate; Drug: Esomeprazole

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan Tablets
  Other Names: TAK-438
  Arms: Vonoprazan 20 mg
Drug: Amoxicillin — Amoxicillin Capsules
Drug: Clarithromycin — Clarithromycin Tablets
Drug: Bismuth Potassium citrate — Bismuth Potassium citrate
Drug: Esomeprazole — Esomeprazole Tablets
  Arms: Esomeprazole 20 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy of helicobacter pylori (HP) eradication with bismuth-containing quadruple therapy with vonoprazan versus esomeprazole in all HP-positive participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called vonoprazan (TAK-438). Vonoprazan is being tested to treat people who have helicobacter pylori infection.

The study is planned to enroll 425 patients at the beginning and will enroll a maximum of approximately 510 patients based on the interim analysis results. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

Vonoprazan 20 mg

Esomeprazole 20 mg

All participants will be asked to take one tablet in combination with bismuth containing quadruple therapy (amoxicillin, clarithromycin and bismuth potassium citrate) twice at the same time each day throughout the study.

This multi-center trial will be conducted in China. The overall time to participate in this study is 10 weeks. Participants will make multiple visits to the clinic, and 28 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Helicobacter pylori (HP)-positive participants as determined by ^13C-urea breath test (^13C-UBT) at the start of the study (Visit 1 [screening]) and who require HP eradication in Physician judgment.

Exclusion Criteria:

1. Participant had any of the following conditions at the start of the study (Visit 1, screening): acute upper gastrointestinal bleeding, active gastric ulcer (GU) or duodenal ulcer (DU) characterized by defective mucos with white coating (with or without adherent blood clots) 3 mm or more in size, acute gastric mucosal lesion (AGML), or acute duodenal mucosal lesion (ADML). However, participants with gastritis, gastric or duodenal erosion are permitted to participate.
2. Participants with Zollinger-Ellison syndrome or gastric acid hypersecretion or those with a history of gastric acid hypersecretion.
3. Participant has a history of malignancy or was treated for malignancy within 5 years before the start of the screening visit (the participant may be included in the study if he/she has cured cutaneous basal cell carcinoma or cervical carcinoma in situ).
4. Participant has a known acquired immunodeficiency syndrome or hepatitis infection, including hepatitis virus carriers (hepatitis B surface antigen [HBsAg] or hepatitis C virus [HCV]- antibody-positive).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Clinical Science, Study Director — Takeda
Locations (29):
- China (29):
  - Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Fuzhou General Hospital of Nanjing Military Command, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Haikou people's Hosptial, Haikou, Hainan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Digestive Department, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University Digestive Department, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Song Z, Du Q, Zhang G, Zhang Z, Liu F, Lu N, Gu L, Kuroda S, Zhou L. Vonoprazan-based quadruple therapy is non-inferior to esomeprazole-based quadruple therapy for Helicobacter pylori eradication: A multicenter, double-blind, randomized, phase 3 study. Chin Med J (Engl). 2025 Nov 20;138(22):2938-2946. doi: 10.1097/CM9.0000000000003437. Epub 2025 Feb 18. PMID 39965795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 29 investigative sites in China from 30 April 2020 to 25 November 2021.
Pre-assignment Details: Helicobacter pylori (HP) positive participants were enrolled and randomized to one of the two treatment groups to either receive quadruple therapy with amoxicillin, clarithromycin, bismuth, and vonoprazan versus quadruple therapy with amoxicillin, clarithromycin, bismuth, and esomeprazole.
Groups:
- Vonoprazan 20 mg: Vonoprazan 20 mg, tablets, orally, twice daily (BID) given in combination with bismuth-containing quadruple therapy (amoxicillin 1 g capsules, clarithromycin 500 mg tablets, and bismuth potassium citrate 600 mg capsules) orally, BID for 2 weeks.
- Esomeprazole 20 mg: Esomeprazole 20 mg, tablets, orally, BID given in combination with bismuth-containing quadruple therapy (amoxicillin 1 g capsules, clarithromycin 500 mg tablets, and bismuth potassium citrate 600 mg capsules) orally, BID for 2 weeks.
Period: Overall Study
Arm/Group | Vonoprazan 20 mg | Esomeprazole 20 mg
Started | 256 | 254
Completed | 254 | 252
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Voluntary Withdrawal by Subject | 0 | 1
Not completed — Reason not Specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of the study drug.
Groups:
- Vonoprazan 20 mg: Vonoprazan 20 mg, tablets, orally, BID given in combination with bismuth-containing quadruple therapy (amoxicillin 1 g capsules, clarithromycin 500 mg tablets, and bismuth potassium citrate 600 mg capsules) orally, BID for 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Vonoprazan 20 mg | Esomeprazole 20 mg | Total
Number analyzed (Participants) | 256 | 254 | 510
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (12.29) | 38.3 (12.13) | 38.9 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 164 | 315
  Male | 105 | 90 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 256 | 254 | 510
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 256 | 254 | 510
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 256 | 254 | 510
Height [Mean (Standard Deviation); unit: cm] | 164.9 (8.23) | 164.3 (7.70) | 164.6 (7.97)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed includes all participants in the FAS who had evaluable data at Baseline, defined as last observation up to Study Day 1.
  kg
    number analyzed (Participants) | 253 | 249 | 502
    (all) | 61.90 (10.579) | 61.15 (9.568) | 61.53 (10.087)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=body weight (kg)/[height (m)^2] Population: Number analyzed includes all participants in the FAS who had evaluable data at Baseline, defined as last observation up to Study Day 1.
  kg/m^2
    number analyzed (Participants) | 253 | 249 | 502
    (all) | 22.66 (2.913) | 22.61 (2.735) | 22.63 (2.823)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Helicobacter Pylori Positive (HP+) Participants With Successful HP Eradication at Week 4 Post-Treatment
Description: HP infection status was determined by ^13C Urea Breath Test (^13C-UBT). The urea breath test is used to detect infection with HP, a bacteria associated with stomach ulcers, by testing individual breath samples in a central laboratory. The percentages are rounded off to report the nearest ten.
Time Frame: Week 4 post-treatment
Population: FAS included all randomized participants who received at least 1 dose of the study drug. Overall number analyzed are the number of participants who had available HP eradication status determined by ^13C-UBT at Week 4 post-treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Vonoprazan 20 mg | Esomeprazole 20 mg
Number analyzed (Participants) | 242 | 240
percentage of participants | 86.8 | 86.7
Statistical Analysis 1: Comparison: Vonoprazan 20 mg vs Esomeprazole 20 mg; Test type: Non-Inferiority — Noninferiority of vonoprazan to esomeprazole was evaluated by Farrington and Manning test using a noninferiority margin of 10% for analysis; p = 0.0009, Farrington and Manning Test; Difference in Proportions = 0.1, 95% CI 2-sided [-5.95 to 6.17] — Difference in proportions for vonoprazan versus esomeprazole was analyzed and the 2-sided Wald confidence interval was used for determining the 95% confidence interval

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to approximately 6 weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Vonoprazan 20 mg | Esomeprazole 20 mg
All-Cause Mortality (participants affected / at risk) | 0/256 | 0/254
Serious Adverse Events (participants affected / at risk) | 3/256 | 5/254
Other Adverse Events (participants affected / at risk) | 110/256 | 91/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Vonoprazan 20 mg (N=256) | Esomeprazole 20 mg (N=254)
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/151 | 0/164 — Number of participants at risk represents the female population in this study.
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0/151 | 1/164 — Number of participants at risk represents the female population in this study.
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0/151 | 1/164 — Number of participants at risk represents the female population in this study.
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 20 mg (N=256) | Esomeprazole 20 mg (N=254)
Faeces discoloured (Gastrointestinal disorders) | 13 | 8
Hepatic function abnormal (Hepatobiliary disorders) | 17 | 9
Protein urine present (Investigations) | 18 | 15
Dysgeusia (Nervous system disorders) | 83 | 74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT04198363/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT04198363/SAP_001.pdf